CLINICAL TRIAL: NCT07217093
Title: Teleconsultation Approach to CTD-ILD Care Delivery in Rural UnderServed CommuniTies (TRUST Initiative)
Status: Not yet recruiting | Type: Observational
Sponsor: St. Lawrence Health System (Other)
Responsible Party: Sponsor
Other Study IDs: EK-TRUST-01
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Interstitial Lung Disease Due to Systemic Disease (Disorder); Interstitial Lung Disease in Patients With Rheumatoid Arthritis; Interstitial Lung Disease Due to Systemic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teleconsultation Group: Patients will receive coordinated care with a regional rheumatologist, regional pulmonologist, and a teleconsultation with an interstitial lung disease specialist from Mayo Clinic

SUMMARY:
Connective tissue disease-associated interstitial lung disease (CTD-ILD) is a rare and complex condition that affects some individuals with autoimmune disorders such as rheumatoid arthritis (RA). It can lead to inflammation and progressive scarring of the lungs, significantly affecting quality of life and overall prognosis.1 Current clinical guidelines recommend that patients with CTD-ILD receive care at specialized academic medical centers with multi-disciplinary teams experienced in managing interstitial lung disease (ILD).2 These centers, however, are often located in urban areas, making access particularly challenging for patients living in rural and underserved regions. In rural, medically underserved areas, the nearest ILD centers can be three or more hours away, posing substantial barriers to timely, consistent, and expert care. These logistical constraints make it difficult for patients residing in rural areas to access the high-quality, specialized care required to manage CTD-ILD effectively.

The Teleconsultation Approach to CTD-ILD Care Delivery in Rural Underserved Communities (TRUST Initiative) it looking to address this gap in access to specialized care. The TRUST Initiative aims to evaluate whether integrating teleconsultation into a personalized, multidisciplinary care model, through regular, structured teleconsultation visits, can enhance the quality and coordination of treatment for patients and potentially other rural underserved patient populations. This model utilizes a regional rheumatologist, a regional pulmonologist and, an interstitial lung disease (ILD) specialist at the Mayo Clinic in Rochester, Minnesota.

This model seeks to overcome the geographic and logistical challenges that prevent patients from accessing specialty care. It also offers a replicable care model for managing other complex chronic diseases in underserved rural communities by leveraging collaborative care, virtual health technology, and structured communication workflows. The study will not only track clinical outcomes such as pulmonary function but also evaluate patient satisfaction, highlighting both the effectiveness and acceptability of this care model.

By addressing disparities in access to specialty care, the TRUST Initiative aims to inform future healthcare delivery strategies for rare and complex diseases in rural and underserved settings nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults aged 18 years or older.
2. Diagnosis and Stable Condition:

   * Confirmed diagnosis of connective tissue disease-associated interstitial lung disease (CTD-ILD) by a physician based on clinical, radiographic, and/or pathological criteria. CTDs may include scleroderma, systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, Sjogren's disease (primary or secondary), inflammatory myopathy including but not limited to dermatomyositis and polymyositis, or any overlap syndrome including one or more of these diseases.
   * Diagnosis of CTD-ILD established at least one year prior to enrollment
3. Residence:

   * Full time resident (at least six months per year) of one of the seven counties of the North Country region of New York (St. Lawrence, Franklin, Jefferson, Lewis, Hamilton, Clinton, Essex)
4. Active Care Relationship:

   * Documented diagnosis of CTD-ILD via any of the following:

     o SLH-affiliated clinician

     o Historical records
     * Determination by PI
   * Or an active SLH medical record (≥1 clinical encounter, test, or treatment in past 24 months)
5. Pulmonary Function Testing and safety labs:

   * Ability and willingness to perform pulmonary function and safety lab tests at local facilities as required by the study protocol.
   * Most recent PFT within 24 months prior to baseline
6. Consent:

   * Provide written informed consent to participate in the study, including consent for data collection and telehealth consultations.

8. Contraception

- Female patients of child-bearing potential (FOCBP) must use at least one highly effective method of contraception between weeks 0 and 48 of the study (complete abstinence, estrogen+progesterone oral contraceptive pill (OCP), progestin-only pill (POP), estrogen+progesterone patch, vaginal ring, Nexplanon, DepoProvera, IUD, bilateral tubal ligation, male partner vasectomy completed at least six months prior to Day 0).

These inclusion criteria ensure that participants are appropriately diagnosed and can engage fully with the teleconsultation-based care model while addressing the program's focus on improving access for rural and other under-resourced populations.

Exclusion Criteria:

1. Severe Cognitive or Mental Health Impairment:

* Individuals with severe cognitive dysfunction or mental health conditions that, in the judgment of the PI, would interfere with the ability to provide informed consent or participate in teleconsultation sessions.

  2. Life Expectancy < 6 Months:
* Participants with a life expectancy of less than six months due to any cause, as determined by the PI.

  3. Other Severe Pulmonary Diseases:
* Individuals with other severe pulmonary conditions determined by PI with input from Sub-Is (e.g., chronic obstructive pulmonary disease [COPD], pulmonary fibrosis unrelated to CTD-ILD, or active lung cancer) that may confound the assessment of CTD-ILD progression.

  4. Inability to Perform Pulmonary Function Tests:
* Participants who are unable to perform or complete the required pulmonary function tests because of physical limitations (e.g., significant respiratory distress or severe disability) or non-compliance.

  5. Active Participation in another Clinical Trial:
* Individuals currently participating in another interventional clinical trial for CTD-ILD or other chronic lung diseases that could interfere with the study outcomes.

  6. Significant Non-Compliance Risk:
* Participants who, in the judgment of the PI, are unlikely to comply with the study protocol or follow-up requirements (e.g., inability to attend teleconsultations, failure to complete pulmonary function tests, or non-adherence to study treatment regimen).

  7. Current ILD Treatment:
* Participants who are currently receiving treatment by an ILD specialist at an ILD center at an academic medical center are not eligible to participate in this study.

  8. Pregnancy or Breastfeeding:
* Pregnant or breastfeeding women.

These exclusion criteria are designed to ensure participant safety, minimize confounding factors, and ensure that participants are able to fully engage in the teleconsultation model and comply with study protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 10 patients diagnosed with CTD-ILD who reside in the rural North Country region of New York.
  For the purpose of this study counties being, but not limited to, St. Lawrence, Franklin, Jefferson, Lewis, Hamilton, Clinton, and Essex counties.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 12 months
  a. Scores from a patient satisfaction survey to assess the perceived quality of teleconsultations-based care including assessments of quality and access to care, cost, and timesaving related to the teleconsultation model. Conducted at the baseline, 6 month, and 12 month visits.

SECONDARY OUTCOMES:
Healthcare Access Metrics | 12 months
  1. Number and percentage of scheduled teleconsultation visits completed.
  2. Adherence rate of teleconsultation arm against their own historical data
Care Coordination and Clinical Outcomes | 12 months
  a. Frequency and nature of communication between local and teleconsulting providers.
Dyspnea-12 | 12 months
  Annual change in the Dyspnea-12 questionnaire (0-36) checked at months 0, 6, and 12
Change in FVC | 12 months
  Annual change in FVC relative to the 24 months prior to enrollment.
Change in DLCO | 12 months
  Annual change in DLCO relative to the 24 months prior to enrollment.
ER Visits | 12 months
  Annual number of ER visits for CTD-ILD exacerbation, with comparison to two years of historical data, teleconsultation arm.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Lawrence Health, Potsdam, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Douthit N, Kiv S, Dwolatzky T, Biswas S. Exposing some important barriers to health care access in the rural USA. Public Health. 2015 Jun;129(6):611-20. doi: 10.1016/j.puhe.2015.04.001. Epub 2015 May 27. PMID 26025176
- [Result] Adegunsoye A, Ryerson CJ. Diagnostic Classification of Interstitial Lung Disease in Clinical Practice. Clin Chest Med. 2021 Jun;42(2):251-261. doi: 10.1016/j.ccm.2021.03.002. PMID 34024401
- See also: Related Info — https://www.thoracic.org/statements/guideline-implementation-tools/diagnosis-of-ipf.php